CLINICAL TRIAL: NCT04985500
Title: Erector Spinae Plane Block vs. Pecto-intercostal Fascial Plane Block vs. Control for Sternotomy: A Prospective Randomized Trial
Brief Title: ESP/PIF for Sternotomy
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Ali Nima Shariat, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY-20-01473
Record Dates: First submitted 2021-07-06; First posted 2021-08-02 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Surgery; Sternotomy
Keywords: ESP Block; PIF Block; Cardiac Surgery; Sternotomy
MeSH Terms: interventions — High-Energy Shock Waves; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Patients will be assigned randomly using a computer-generated table of numbers to one of the three groups: 1) ESP group, 2) PIF group, or 3) no block group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The anesthesiologist assessing the patient will be blinded
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ESP group (Experimental): Patient will receive ESP block with ultrasound guidance the transverse process of the vertebra at T7 is visualized and 20 mL of 0.25% bupivacaine will be injected between the transverse process and the erector spinae muscle on each side using a 21-gauge block needle.
  Interventions: Procedure: ESP block; Procedure: Ultrasound; Drug: Bupivacain
- PIF group (Experimental): Patient will receive PIF block after intubation with ultrasound placed 1-2 cm lateral to the sternal border and the pectoralis major and external intercostal muscles are visualized at the level of ribs 3-4 where 10 mL of 0.25% bupivacaine will be injected on each side using a 21-gauge block needle.
  Interventions: Procedure: PIF block; Procedure: Ultrasound; Drug: Bupivacain
- No Block group (No Intervention): Patient will not receive block.

INTERVENTIONS:
Procedure: ESP block — peripheral nerve block
  Other Names: erector spinal plane block
  Arms: ESP group
Procedure: PIF block — peripheral nerve block
  Other Names: pecto-intercostal fascial plane block
  Arms: PIF group
Procedure: Ultrasound — Ultrasound guidance
  Arms: ESP group; PIF group
Drug: Bupivacain — 10-20 mL of 0.25% bupivacaine
  Arms: ESP group; PIF group

SUMMARY:
This is a randomized study. The purpose of this study is to evaluate the effect of post-surgical pain control of two types of peripheral nerve blocks, specifically erector spinal plane (ESP) block and pecto-intercostal fascial (PIF) plane block.

90 subjects, from 18-85 years of age, undergoing cardiac surgery with median sternal incision will be enrolled at Mount Sinai Morningside Hospital Center. Study participation will last from the time of pre-operative evaluation to 72 hours after surgery. Subjects will be randomly assigned to receive 1 of the 3 different regimens at the beginning of surgery. Opioid consumption and pain scores after surgery will be evaluated. Though unlikely, risks include systemic absorption of local anesthetic, which can result in both central nervous system and cardiac toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-85 years old
* Scheduled to undergo cardiac procedures involving sternotomy
* All genders

Exclusion Criteria:

* ASA class V
* Urgent or emergent surgery
* Contraindications to administration of local anesthesia (e.g. local anesthetic allergy)
* History of substance abuse or chronic opioid use
* Patient refusal or inability to consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Opioid Consumption during first 24 hours post-op | Post-operative 24 hours
  The amount of opioid consumption (in mg IV morphine equivalents) during the first 24 hours post-op in patients undergoing cardiac surgeries with median sternotomy.
Opioid Consumption during first 48 hours post-op | Post-operative 48 hours
  The amount of opioid consumption (in mg IV morphine equivalents) during the first 48 hours post-op in patients undergoing cardiac surgeries with median sternotomy.
Opioid Consumption during first 72 hours post-op | Post-operative 72 hours
  The amount of opioid consumption (in mg IV morphine equivalents) during the first 72 hours post-op in patients undergoing cardiac surgeries with median sternotomy.

SECONDARY OUTCOMES:
Visual Analogue Score (VAS) Pain Score post-op 24 hours | Post-operative 24 hours
  VAS Pain Score from 0-10, with higher score indicating more pain. The average VAS pain scores during the first 24 hours post-op in patients undergoing cardiac surgeries with median sternotomy.
Visual Analogue Score (VAS) Pain Score post-op 48 hours | Post-operative 48 hours
  VAS Pain Score from 0-10, with higher score indicating more pain. The average VAS pain scores during the first 48 hours post-op in patients undergoing cardiac surgeries with median sternotomy.
Visual Analogue Score (VAS) Pain Score post-op 72 hours | Post-operative 72 hours
  VAS Pain Score from 0-10, with higher score indicating more pain. The average VAS pain scores during the first 72 hours post-op in patients undergoing cardiac surgeries with median sternotomy.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Shariat, M.D., Principal Investigator — Mount Sinai West and Morningside Hospitals; Himani Bhatt, D.O., Study Director — Mount Sinai West and Morningside Hospitals; Shenghao Fang, M.D., Study Director — Mount Sinai West and Morningside Hospitals
Locations (1):
- Mount Sinai Morningside Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No